CLINICAL TRIAL: NCT02957656
Title: A Phase I Study In Healthy Adults To Assess The Safety And Immunogenicity Of Priming With Live Attenuated A/H7N9 Influenza Virus Vaccine Followed By Inactivated A/H7N9 Influenza Virus Vaccine With AS03 Adjuvant
Brief Title: Safety and Immunogenicity of Priming With Live Attenuated A/H7N9 Influenza Virus Vaccine Followed By Inactivated A/H7N9 Influenza Virus Vaccine With AS03 Adjuvant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-002
Record Dates: First submitted 2016-11-02; First posted 2016-11-08 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Influenza A Virus, H7N9 Subtype
MeSH Terms: interventions — AS03 adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1: H7N9 pLAIV + AS03-adjuvanted H7N9 pIIV (Experimental): Participants will receive one dose of approximately 10^7.0 FFU of H7N9 pLAIV at study entry (Day 0). They will receive one dose of 15 µg of AS03-adjuvanted H7N9 pIIV at Day 84.
  Interventions: Biological: H7N9 pLAIV; Biological: H7N9 pIIV; Biological: AS03 adjuvant
- Group 2: AS03-adjuvanted H7N9 pIIV + AS03-adjuvanted H7N9 pIIV (Experimental): Participants will receive one dose of 15 µg of AS03-adjuvanted H7N9 pIIV at study entry (Day 0) and one dose of 15 µg of AS03-adjuvanted H7N9 pIIV at Day 84.
  Interventions: Biological: H7N9 pIIV; Biological: AS03 adjuvant
- Group 3: AS03-adjuvanted H7N9 pIIV (Experimental): Participants will receive one dose of 15 µg of AS03-adjuvanted H7N9 pIIV at study entry (Day 0).
  Interventions: Biological: H7N9 pIIV; Biological: AS03 adjuvant
- University of Rochester URMC 13-001 Participants (Experimental): Participants received one dose of 10^7 FFU of H7N9 pLAIV at study entry (Day 0), one dose of 10^7 FFU of H7N9 pLAIV at Day 28, and one dose of 30 µg of unadjuvanted H7N9 pIIV at Day 84.
  Interventions: Biological: H7N9 pLAIV; Biological: H7N9 pIIV
- Johns Hopkins School of Public Health CIR293 Participants (Experimental): Participants received one dose of 10^7 FFU of H7N9 pLAIV at study entry (Day 0), one dose of 10^7 FFU of H7N9 pLAIV at Day 28, and one dose of 30 µg of unadjuvanted H7N9 pIIV at Day 84.
  Interventions: Biological: H7N9 pLAIV; Biological: H7N9 pIIV

INTERVENTIONS:
Biological: H7N9 pLAIV — 10^7.0 fluorescent focus units (FFU); delivered by an Accuspray device
  Other Names: Live Influenza A Vaccine H7N9 (6-2) AA ca Recombinant (A/Anhui/1/2013 (H7N9) x A/Ann Arbor/6/60 ca)
  Arms: Group 1: H7N9 pLAIV + AS03-adjuvanted H7N9 pIIV; Johns Hopkins School of Public Health CIR293 Participants; University of Rochester URMC 13-001 Participants
Biological: H7N9 pIIV — Administered by intramuscular injection in the deltoid.
Biological: AS03 adjuvant — Mixed with H7N9 pIIV vaccine; administered by intramuscular injection in the deltoid
  Arms: Group 1: H7N9 pLAIV + AS03-adjuvanted H7N9 pIIV; Group 2: AS03-adjuvanted H7N9 pIIV + AS03-adjuvanted H7N9 pIIV; Group 3: AS03-adjuvanted H7N9 pIIV

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of one dose of H7N9 pandemic live attenuated influenza vaccine (H7N9 pLAIV) followed by AS03-adjuvanted H7N9 pandemic inactivated influenza vaccine (H7N9 pIIV).

DETAILED DESCRIPTION:
This study will evaluate the safety and immunogenicity of one dose of H7N9 pandemic live attenuated influenza vaccine (H7N9 pLAIV) followed by AS03-adjuvanted H7N9 pandemic inactivated influenza vaccine (H7N9 pIIV).

This study will enroll healthy adults who will choose which study group to join. Participants in Group 1 will receive one dose of H7N9 pLAIV in an inpatient setting at study entry (Day 0). They will remain in an isolation unit through at least Day 9. They will also receive one dose of AS03-adjuvanted H7N9 pIIV on Day 84.

Participants in Group 2 will receive one dose of AS03-adjuvanted H7N9 pIIV at study entry (Day 0) and a second dose of AS03-adjuvanted H7N9 pIIV at Day 84. Participants in Group 3 will receive one dose of AS03-adjuvanted H7N9 pIIV at study entry (Day 0).

All participants will attend multiple study visits through Day 264. Study visits may include blood collection, physical examinations, and nasal wash and nasal wick procedures.

These three groups will be compared to two historical control groups who received one dose of H7N9 pLAIV at study entry (Day 0), one dose of H7N9 pLAIV at Day 28, and one dose of unadjuvanted H7N9 pIIV at Day 84.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant, non-breastfeeding females between 20 years and 49 years of age, inclusive. Children will not be recruited or enrolled in this study because they are not in the apparent risk group, for safety considerations, and because of the need for isolation.
* Are in good health, as determined by medical history and targeted physical examination to ensure any existing medical diagnoses or conditions (except those exclusionary) are stable. More information on this criterion can be found in the protocol.
* Agree to storage of blood specimens for future research.
* Available for the duration of the trial. Subjects must be willing and able to remain within the Isolation Unit for the specified duration of confinement.
* Provide written informed consent prior to initiation of any study procedures, including future use of specimens.
* Female subjects of childbearing potential must agree to use effective birth control methods for the duration of the study (for example, pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; intrauterine device; abstinence from heterosexual intercourse, surgical sterilization). All female subjects will be considered being of childbearing potential except those who have undergone hysterectomy or tubal ligation and those in whom menopause occurred at least 1 year prior to the study.
* Agrees not to participate in another clinical trial with an investigational product for the entire duration of the study.
* Oral temperature is less than 100.4°F.
* Pulse is 50 to 115 bpm, inclusive.
* Systolic blood pressure is 85 to 150 mm Hg, inclusive.
* Diastolic blood pressure is 55 to 95 mm Hg, inclusive.
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination.

Exclusion Criteria:

* Pregnancy as determined by a positive human choriogonadotropin (beta-HCG) test.
* Currently breastfeeding or planning to breastfeed at some point during the duration of the study.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, electrocardiogram (EKG) and/or laboratory studies including urine testing. Alanine aminotransferase (ALT) levels greater than 2 times the upper normal limit will be exclusionary at baseline, prior to vaccination.
* Any current illness requiring daily medication other than the following: vitamins, birth control, anti-hypertensive medication, antihistamines, anti-depressant medication, cholesterol-lowering medication, treatment for gastroesophageal reflux disease, and thyroid medication unless approved by the PI.
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
* Previous enrollment in an H7 or H9 influenza vaccine trial or in any study of an avian influenza vaccine.
* Seropositive to the H7N9 influenza A virus (serum HAI titer greater than 1:8).
* Positive urine drug toxicology test indicating narcotic use/dependency.
* Have medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
* Have a history of severe reactions following previous immunization with licensed or unlicensed influenza virus vaccines.
* Have known hypersensitivity or allergy to eggs, egg or chicken protein, squalene-based adjuvants, or other components of the study vaccine.
* Allergy to oseltamivir as determined by subject report.
* Current diagnosis of asthma or reactive airway disease (within the past 2 years).
* History of Guillain-Barré Syndrome.
* Positive enzyme-linked immunosorbent assay (ELISA) and confirmatory Western blot tests for human immunodeficiency virus-1 (HIV-1).
* Positive ELISA and confirmatory test (e.g., recombinant immunoblot assay) for hepatitis C virus (HCV).
* Positive hepatitis B virus surface antigen (HBsAg) by ELISA.
* Known immunodeficiency syndrome.
* Use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to vaccination.
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study vaccination.
* Planned receipt of any vaccine from the first study vaccination through the follow-up visit at approximately 180 days after the final study vaccination.
* History of asplenia.
* Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 36 months prior to vaccination.
* Have known active neoplastic disease or a history of any hematologic malignancy.
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination.
* Current smoker unwilling to stop smoking for the duration of the inpatient stay.

  * A current smoker includes anyone stating they currently smoke or use any amount of a tobacco product, including electronic cigarettes.
  * After admission to the unit, nicotine patches will be provided to current smokers who request them for the inpatient portion of the study.
* Travel to the Southern Hemisphere within 14 days prior to study vaccination.
* Travel on a cruise ship within 14 days prior to study vaccination.
* Receipt of another investigational vaccine or drug within 30 days prior to study vaccination.
* Any potential Immune Mediated Disease (pIMD) listed in the protocol, or other diseases that may have an autoimmune origin.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Rates of local and systemic reactogenicity events | Measured through Day 264
Development of adverse events at any time point during the study | Measured through Day 264
Geometric mean titer (GMT) of H7N9-specific serum hemagglutination inhibition (HAI) and/or microneutralization (MN) antibody responses | Measured through Day 264
Rates of H7N9-specific serum HAI and/or MN antibody responses | Measured through Day 264

CONTACTS AND LOCATIONS:
Overall Officials: Angela Branche, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States